CLINICAL TRIAL: NCT04355156
Title: A Phase II Double Blind, Randomised Controlled Trial of VEGF Inhibitor Axitinib Monotherapy With Early Dynamic Contrast Enhanced Ultrasound Monitoring in Chemorefractory Third Line Metastatic Colorectal Cancer
Brief Title: Axitinib Monotherapy With Early Dynamic Contrast Enhanced Ultrasound Monitoring in Chemorefractory Third Line Metastatic Colorectal Cancer
Acronym: AXMUS-C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WS913975; 2011-002598-49 (EudraCT Number)
Record Dates: First submitted 2020-04-15; First posted 2020-04-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Axitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Axitinib (Experimental): small molecule multi-kinase inhibitor
  Interventions: Drug: Axitinib
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Axitinib — * All patients randomised to this arm will receive 3mg BD, and increased at 2 weeks to 5mg BD
  * Outpatient monitoring at 2 week intervals for a minimum of 8 weeks, with 2 weekly liver contrast ultrasound for assessment of differential blood supply (CEHPI)
  * At 8 weeks, after tumour CT RECIST assessments, responders will continue monotherapy. In non-responders, those with disease progression, monotherapy can be continued if patient chooses to continue and if tolerated
  Arms: Axitinib
Drug: Placebo — * All patients receiving placebo will receive tablets to take BD
  * Outpatient monitoring at 2 week intervals for a minimum of 8 weeks, with 2 weekly liver contrast ultrasound for assessment of differential blood supply (CEHPI)
  Arms: Placebo

SUMMARY:
This is a study of Axitinib versus placebo as monotherapy for people with colorectal cancer who have liver metastases and who have relapsed within 6 months of their last chemotherapy regime. The research will also look at the potential of CEHPI (Contrast Enhanced Hepatic Perfusion Index) reduction, a technique developed for this research to measure the changes in how the blood vessels pump blood into the different liver metastases (tumours) and therefore to assess and predict response to treatment.

DETAILED DESCRIPTION:
Colorectal cancer is the second most common cause of cancer death in the UK with an average 5-year survival of 50%. There is a lack of classical chemotherapy response in metastatic colorectal cancer with the approved drugs currently on the market, which has prompted the investigation of angiogenesis inhibitors as a new chemotherapeutic agent. Pre-clinical use of angiogenesis inhibitors with conventional cytotoxic chemotherapy has shown to have more effect, but so far these results have not been replicated in human studies. Furthermore, the toxicity profiles for these drugs when combined with chemotherapy has so far outweighed any benefit they may hold for patients. With this in mind, are we perhaps not dosing correctly? Would changing the dosing schedule optimise the balance between efficacy versus toxicity?

AXMUS-C is a phase II randomised, placebo-controlled study testing the efficacy of the VEGF inhibitor, Axitinib, as monotherapy for patients with chemo-refractory colorectal cancer with liver metastases.

A-013736 (Axitinib) is a selective inhibitor of vascular endothelial growth factor (VEGF) receptors 1, 2 and 3, and is therefore classed as an angiogenesis inhibitor with VEGF receptors effectively being blocked and thus cannot stimulate the signalling pathway responsible for cell proliferation resulting in the growth of blood vessels to feed the tumour. Several studies in other solid tumours have shown that when taken orally the main side effect of Axitinib is fatigue, with 51% of subjects reporting varying grades of severity. Axitinib has been approved by the U.S. Food and Drug Administration (FDA) for the treatment of advanced renal cell carcinoma after failure of one prior systemic therapy. It has not been approved for colorectal cancer.

Additionally, the research will also assess the potential for early CEHPI (Contrast Enhanced Hepatic Perfusion Index) reduction to predict response to therapy with Axitinib, with the hypothesis being that patients with an early ≥20% reduction in CEHPI will have improved overall survival, compared to those who do not. Early relative reductions of over 20% has previously been shown to correlate with conventional stable disease and partial response by RECIST. [CEHPI] has been developed with the idea that it can identify responders to the anti-VEGF therapy much earlier than the conventionally used established RECIST method. It is a technique that measures the changes in how the blood vessels pump blood into the different liver metastases (tumours) and therefore can be used to assess and predict response to treatment, as it is known that arterialisation support the growth of malignant tumours in the liver whereas usually the portal vein supplies 70% of the blood to normal liver parenchyma. Contrast enhanced ultrasound differ from the standard ultrasound with the intravenous injection of 2mL of SonoVue before the Philips iu22 platform and a C5-1 transducer are used to record a one-minute cine loop.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria to be eligible for enrolment into the study:

* Histologically or cytologically confirmed adenocarcinoma of the colon or rectum with liver metastas(es). At least one of which should not have had any focal therapy including radiofrequency ablation, chemoembolization, ethanol or cryoablation.
* Failed at least 2 chemotherapy regimens in advanced disease.
* Evidence of unidimensionally measurable disease as defined by the Response Evaluation Criteria in Solid Tumors (RECIST).
* 18 years of age or older.
* ECOG performance status of 0 or 1.
* Resolution of all acute toxic effects of prior therapy e.g. radiotherapy or surgical procedure to NCI CTCv4 grade ≤1.
* Adequate organ function as defined by the following criteria:

Serum aspartate aminotransferase (AST; serum glutamic oxaloacetic transaminase [SGOT]) and serum alanine aminotransferase (ALT; serum glutamic pyruvic transaminase [SGPT]) ≤2.5 x upper limit of normal (ULN). For patients with liver metastases, <5 x ULN.

Total serum bilirubin <1.5 x ULN Serum albumin ≥3.0 g/dL Absolute neutrophil count ≥1500/µL Platelets ≥100,000/µL Haemoglobin ≥9.0 g/dL Serum creatinine ≤1.5 x ULN

* Signed and dated informed consent form
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures, including the completion of patient reported outcome measures.
* At least 2 weeks since the end of prior systemic treatment (4 weeks for Bevacizumab-containing regimens), radiotherapy, or surgical procedure with resolution of all treatment-related toxicity to NCI CTCAE Version 3.0 grade ≤1 or back to baseline except for alopecia or hypothyroidism.
* No evidence of pre-existing uncontrolled hypertension as documented by 2 baseline blood pressure readings taken at least 1 hour apart. The baseline systolic blood pressure readings must be ≤140 mm Hg, and the baseline diastolic blood pressure readings must be ≤90 mm Hg. Patients whose hypertension is controlled by antihypertensive therapies are eligible.
* Women of childbearing potential must have a negative serum or urine pregnancy test within 3 days prior to treatment.
* Signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to enrolment.

Exclusion Criteria:

The presence of any of the following will exclude a patient from enrolment:

* Non-exposed to both oxaliplatin and irinotecan FP based cytotoxic chemotherapy (prior pelvic radiation therapy including adjuvant or neoadjuvant chemo-radiation therapy for resected rectal cancer is allowed provided it is completed within 4 weeks prior to study entry)
* Less than 6 months from completion of adjuvant chemotherapy to diagnosis or documentation of recurrent cancer
* Palliative radiotherapy to non-target, metastatic lesions will be allowed provided it was completed within 4 weeks prior to study entry.
* Prior surgery or IMP within 4 weeks prior to study entry
* Current treatment within another therapeutic clinical trial.
* Presence of grade ≥2 peripheral neuropathy.
* Known dihydropyrimidine dehydrogenase deficiency or severe hypersensitivity reaction to 5-FU
* Grade ≥2 thrombocytopenia (i.e., platelet count <75,000/µL), grade 3 neutropenia (i.e., absolute neutrophil count <1000/µL), or grade 3 non-hematologic adverse event associated with prior adjuvant oxaliplatin and/or 5-FU treatment.
* History of significant bleeding within the past 3 months, including gross haemoptysis or haematuria, or underlying coagulopathy.
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study enrolment, unless affected area has been removed surgically.
* On-going cardiac dysrhythmias of grade ≥2, atrial fibrillation of any grade, or QTc interval to >450 msec for males and >470 msec for females.
* Hypertension uncontrolled by medication (>150/100 mmHg despite optimal medical therapy).
* On-going treatment with therapeutic doses of warfarin (however, low dose warfarin up to 2mg daily for deep vein thrombosis prophylaxis is allowed). Low molecular weight heparin (LMWH) is allowed.
* Diagnosis of any second malignancy within the last 3 years that is potentially liable to interfere with study outcomes (basal cell carcinoma, squamous cell skin cancer, or in situ carcinoma and hormone controlled locally advanced prostate cancer that has been adequately treated with no evidence of recurrent disease for 12 months, are allowed)
* History of or known brain metastases, spinal cord compression, or carcinomatous meningitis, or new evidence of brain or leptomeningeal disease on screening CT or MRI scan.
* Any of the following within the 12 months prior to study drug administration: severe/unstable angina, myocardial infarction, symptomatic congestive heart failure, cerebrovascular accident, or transient ischemic attack.
* Known human immunodeficiency virus (HIV) infection.
* Pregnancy, breastfeeding, or unwillingness/inability to employ an effective method of birth control/contraception to prevent pregnancy during treatment and for up to 3 months after discontinuing study drug if of reproductive potential.
* Other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that would impart, in the judgement of the investigator, excess risk associated with study participation or study drug administration, or which, in the judgment of the investigator would make the patient inappropriate for entry into the trial.
* Non-English speaking
* Major surgery <4 weeks or radiation therapy <2 weeks of starting the study treatment. Prior palliative radiotherapy to metastatic lesion(s) is permitted, provided there is at least one measurable lesion that has not been irradiated.
* Gastrointestinal abnormalities including: inability to take oral medication; requirement for intravenous alimentation; prior surgical procedures affecting absorption including total gastric resection; treatment for active peptic ulcer disease in the past 6 months; active gastrointestinal bleeding, unrelated to cancer, as evidenced by hematemesis or melaena in the past 3 months without evidence of resolution documented by endoscopy or colonoscopy; malabsorption syndromes
* Current use or anticipated need for treatment with drugs that are known potent CYP3A4 inhibitors (ie, grapefruit juice, verapamil, ketoconazole, miconazole, itraconazole, erythromycin, telithromycin, clarithromycin, indinavir, saquinavir, ritonavir, nelfinavir, lopinavir, atazanavir, amprenavir, fosamprenavir and delavirdine).
* Current use or anticipated need for treatment with drugs that are known CYP3A4 or CYP1A2 inducers (ie, carbamazepine, dexamethasone, felbamate, omeprazole, phenobarbital, phenytoin, amobarbital, nevirapine, primidone, rifabutin, rifampin, and St. John's wort).
* Requirement of anticoagulant therapy with oral vitamin K antagonists. Low-dose anticoagulants for maintenance of patency of central venous access devise or prevention of deep venous thrombosis is allowed. Therapeutic use of low molecular weight heparin is allowed.
* Active seizure disorder or evidence of brain metastases, spinal cord compression, or carcinomatous meningitis.
* A serious uncontrolled medical disorder or active infection that would impair their ability to receive study treatment.
* Any of the following within the 12 months prior to study drug administration: myocardial infarction, uncontrolled angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack and 6 months for deep vein thrombosis or pulmonary embolism.
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness.
* History of a malignancy (other than renal cell cancer) except those treated with curative intent for skin cancer (other than melanoma), in-situ breast or in situ cervical cancer, or those treated with curative intent for any other cancer with no evidence of disease for 2 years.
* Dementia or significantly altered mental status that would prohibit the understanding or rendering of informed consent and compliance with the requirements of this protocol.
* Female patients who are pregnant or lactating, or men and women of reproductive potential not willing or not able to employ an effective method of birth control/contraception to prevent pregnancy during treatment and for 6 months after discontinuing study treatment The definition of effective contraception should be in agreement with local regulation and based on the judgment of the principal investigator or a designated associate.
* Other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2012-09-17 (Actual); Primary Completion 2019-02-22 (Actual); Study Completion 2019-02-22 (Actual)

PRIMARY OUTCOMES:
Overall survival | Through study completion, an average of 1 year
  Difference in median overall survival between patients in the Axitinib arm who achieve a reduction in CEHPI index of at least 20% from baseline and those who do not achieve in both Axitinib and placebo arms

SECONDARY OUTCOMES:
Imaging | Through study completion, an average of 1 year
  Comparison of disease progression in patients who fail to display reduction in CEHPI at weeks according to RECIST V1.1
Objective response rate | Through study completion, an average of 1 year
  Best objective response rate in Axitinib versus placebo groups
Objective response rate | Through study completion, an average of 1 year
  Best objective response rate in CEHPI responders versus non-responders
Monitoring of adverse reactions | Through study completion, an average of 1 year
  Adverse events graded by Chemotherapy toxicity criteria (CTC) V4 grading
Progression free survival | Through study completion, an average of 1 year
  Progression free survival and 6 and 9 month survival percentages and 'duration on treatment' between Axitinib and placebo
Progression free survival secondary outcome | Through study completion, an average of 1 year
  Progression free survival and 6 and 9 month survival percentages and 'duration on study treatment' between CEHPI responders and non-responders
Monitoring dose reductions and the reasons behind them | Through study completion, an average of 1 year
  Minimum dose of Axitinib required to reduce CEHPI significantly, in responders and in patients who require dose reductions due to toxicity

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided